CLINICAL TRIAL: NCT02840214
Title: Impact of Transcranial Direct Current Stimulation on Fatigability and Fatigue Induced by a Selective Attention Task
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1035
Record Dates: First submitted 2016-06-27; First posted 2016-07-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- tDCS rescue group (Active Comparator): Subjects assigned to this arm will receive transcranial direct current stimulation (tDCS) that delivers a constant, small current (2 milliAmp) across specific regions of the brain through electrodes placed on the scalp half-way through the 3-hour fatigue task.
  Interventions: Device: transcranial direct current stimulation
- Sham Treatment Group (Placebo Comparator): Subjects assigned to this arm will initially receive current of the same intensity for a period of 30 seconds and then gradually turned off.
  Interventions: Device: sham tDCS
- tDCS prevent group (Active Comparator): Subjects assigned to this arm will receive transcranial direct current stimulation (tDCS) that delivers a constant, small current (2 milliAmp) across specific regions of the brain through electrodes placed on the scalp at the beginning of the task.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Soterix tDCS RCT device given over left DLPFC for 20 minutes at 2mA.
  Other Names: tDCS
  Arms: tDCS prevent group; tDCS rescue group
Device: sham tDCS — Soterix tDCS RCT device given over left DLPFC with 30 second ramp on and off of current
  Other Names: Placebo
  Arms: Sham Treatment Group

SUMMARY:
This research project is focusing on changes in mental fatigue due to transcranial direct current stimulation (tDCS) in healthy individuals. The study aim is to see if mental fatigue can be rescued by administering a safe dose of tDCS. tDCS has been shown to decrease fatigue in healthy individuals experiencing extended wakefulness, and the investigators aim to investigate if similar results can be found in a fatigue inducing task. This is a single-blind randomized control trial that will compare mental fatigue between tDCS treatment and sham treatment groups through both subjective and objective measures. Objective fatigue will be measured by reaction time with the Stroop test and subjective fatigue will be measured by the multidimensional fatigue inventory questionnaire.

DETAILED DESCRIPTION:
Right handed healthy individuals aged 18-40 will be eligible to participate. Participants will be randomized in a 1:1:1 ratio to receive real or placebo 2mA tDCS delivered for 20 minutes while performing a 3 hour computerized cued Stroop task. Groups will receive real or sham stimulation during the first 20 minutes or 90-110 minutes into the task. Groups will be: 1) Sham (sham given at both time points); 2) Prevent (real will be given during first 20 minutes to try to prevent or delay fatigue and sham given at second time point); or 3) Rescue (sham will be given initially and real given at 90-110 minutes to see if performance can be rescued after fatigue has set in). The primary outcome measure will be the slope of change for intra-individual variability of response time for correct items and regression models will be used to determine whether real preventative or rescue tDCS alters the rate of performance change relative to sham stimulation. Accuracy and mean response time will also be examined as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* normal or corrected-normal vision,

Exclusion Criteria:

* pregnant women,
* history of medical conditions associated with fatigue, including, but not limited to:

  * Parkinson's disease,
  * Alzheimer's disease,
  * diabetes mellitus,
  * hypothyroidism,
  * chronic fatigue syndrome,
  * anemia,
  * infectious mononucleosis,
  * irritable bowel syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance fatigability | over 3 hours of a single fatigability task (one time visit study)
  This will be measured by change in intraindividual variability of reaction time from the Stroop Fatigue Paradigm which will be quantified as the rate of change in mean reaction time over 3 hours modeled using linear regression.

SECONDARY OUTCOMES:
Change in perceived fatigue | Baseline then every 30 minutes for 3 hours
  This will be assessed by visual analogue scale of fatigue performed at baseline and every 30 minutes of the task and the slope of change in perceived fatigue modeled using linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Benzi Kluger, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be released to other researchers upon request.